CLINICAL TRIAL: NCT04107662
Title: A Prospective, Multi-Center, Non-Randomized Study to Identify Intracranial Hemorrhage by Using an In-Vitro Device, Tbit™ System
Brief Title: Biomarkers of Traumatic Brain Injury With Tbit System
Status: Not yet recruiting | Type: Observational
Sponsor: BioDirection Inc (Industry)
Responsible Party: Sponsor
Organization: NanoDx (Industry)
Other Study IDs: BDI-TBIT-03
Record Dates: First submitted 2019-09-17; First posted 2019-09-27 (Actual); Last update posted 2024-04-05 (Actual); Status verified 2024-04

CONDITIONS: Brain Injuries, Traumatic
Keywords: brain; injuries; disease; trauma; nervous system; wounds
MeSH Terms: conditions — Brain Injuries, Traumatic; Wounds and Injuries; Disease; Neurologic Manifestations

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

GROUPS / COHORTS (1):
- Traumatic Brain Injury
  Interventions: Device: Tbit system

INTERVENTIONS:
Device: Tbit system — Suspected traumatic brain injury with head CT
  Other Names: Head CT scan and blood draw within 12 hours of injury

SUMMARY:
A prospective, multi-center, non-randomized, pivotal study to assess the safety and efficacy of the Tbit™ System to aid in patient evaluation, suspected of traumatic brain injury, as adjunct companion test to radiologic standard of care, Cranial Computerized Tomography (CCT).

ELIGIBILITY:
Inclusion Criteria:

* At least 18 years of age
* Presents to the Emergency Department with suspected traumatic brain injury
* Prescribed a non-contrast CCT as part of routine emergency care within 24 hours from injury
* Blood sample collected for Tbit™ System within 12 hours of injury
* Willing and able to provide informed consent or obtain consent from legal authorized representative (LAR)

Exclusion Criteria:

* Suspect of ischemic or hemorrhagic stroke with subsequent incidental trauma based on ED examination
* Subject suspect of need of craniotomy for the acute trauma for this event
* External signs compatible with a depressed skull fracture based on ED exam
* Subject requiring administration of blood transfusion after injury and prior to study blood draw
* Subject for whom timing of injury is unable to be estimated within 1 hour of certainty
* Subject with a condition precluding entry into the CT scanner
* Subject who had neurodegenerative disease or other neurological disorder including dementia, Parkinson's disease, multiple sclerosis, seizures, brain tumors, stroke or TIA within the last 30 days, or history of neurosurgery
* Known or suspected to be pregnant
* Prisoner or under incarceration
* Participating in another clinical research study prior to this study completion

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Male and female participants (≥18 years of age) that present to the Emergency Department with suspected non-penetrating blunt trauma within 24 hours from injury and who receive a CT scan as a standard of care.
Sampling Method: Probability Sample
Enrollment: 740 (Estimated)
Dates: Start 2024-12-01 (Estimated); Primary Completion 2025-05-30 (Estimated); Study Completion 2025-05-30 (Estimated)

PRIMARY OUTCOMES:
Cranial CT Intracranial Hemorrhage findings and the binary Tbit™ System (positive/negative) | within 12 hours from injury on day 0 of ED presentation
  Cranial CT Intracranial Hemorrhage findings (positive/negative) and the binary Tbit™ System results (positive/negative) of each sample.
Tbit™ System sensitivity and specificity | within 12 hours from injury on day 0 of ED presentation
  Tbit™ System sensitivity and specificity relative to the standard-of-care (SOC)

SECONDARY OUTCOMES:
Negative predictive value of the Tbit™ System | within 12 hours from injury on day 0 of ED presentation
  Negative predictive value of the Tbit™ System
Positive predictive value of the Tbit™ System | within 12 hours from injury on day 0 of ED presentation
  Positive predictive value of the Tbit™ System
Overall accuracy of the Tbit™ System | within 12 hours from injury on day 0 of ED presentation
  Overall accuracy of the Tbit™ System
Safety and adverse event profile | 6 months
  Safety and adverse event profile

OTHER OUTCOMES:
Tbit™ System User Satisfaction Survey | 6 months
  Tbit™ System User Satisfaction Survey to evaluate the Tbit ease of use by device operators

CONTACTS AND LOCATIONS:
Overall Officials: Jerika Acosta, BSc, Study Director — Medicept Inc.